CLINICAL TRIAL: NCT07194954
Title: Effects of Combined Dietary Fiber and Probiotic Supplementation on Gut Microbiota, Immune Function, and Clinical Outcomes in Patients With Advanced Colorectal Cancer: A Prospective Randomized Controlled Trial
Brief Title: Dietary Fiber and Probiotics in Advanced Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Feifei Wang, Principal Investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022S00116
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer (MSI-H); Malnutrition (Calorie)
MeSH Terms: conditions — Colorectal Neoplasms; Malnutrition | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention Group (Experimental): Patients were randomized to receive standard nutritional support supplemented with a daily combined formulation of dietary fiber and multi-strain probiotics for 12 weeks.
  Interventions: Dietary Supplement: Combined Dietary Fiber and Probiotics.
- Active Comparator: Control Group (Active Comparator): Patients were randomized to receive standard nutritional support alone for 12 weeks.
  Interventions: Other: Standard Nutritional Support

INTERVENTIONS:
Dietary Supplement: Combined Dietary Fiber and Probiotics. — The intervention consisted of a daily oral administration of 20g of a mixed dietary fiber powder (FibroBalance®, containing inulin, pectin, and β-glucan) and one multi-strain probiotic capsule (ProbioCare Forte®, delivering 10^9 CFU of Lactobacillus acidophilus NCFM, Bifidobacterium lactis Bi-07, and Streptococcus thermophilus St-21).
  Arms: Experimental: Intervention Group
Other: Standard Nutritional Support — This included dietary counseling from a registered dietitian and, if necessary, a standard oral nutritional supplement (Ensure®) to meet estimated energy and protein requirements.
  Arms: Active Comparator: Control Group

SUMMARY:
This single-center, prospective, randomized controlled trial was conducted to evaluate the efficacy of a 12-week combined dietary fiber and probiotic supplementation on gut microbiota, immune function, nutritional status, and survival outcomes in malnourished patients with advanced colorectal cancer undergoing conventional therapy, compared to standard nutritional support alone.

DETAILED DESCRIPTION:
Patients with advanced colorectal cancer often suffer from malnutrition and immune suppression, which can negatively impact treatment outcomes. This study investigated whether modulating the gut microbiota could improve clinical outcomes. A total of 80 eligible patients were randomly assigned in a 1:1 ratio to an intervention group or a control group. The intervention group (n=40) received standard nutritional support plus a daily supplement of mixed dietary fiber and multi-strain probiotics for 12 weeks. The control group (n=40) received standard nutritional support alone. Key endpoints, including immune markers (IgA, IgG, CD4+/CD8+ ratio), gut microbiota composition (16S rRNA sequencing), nutritional status (BMI, PG-SGA), and quality of life (WHOQOL-100), were assessed at baseline and after 12 weeks. Survival was monitored for 18 months to determine the impact on short-term prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of stage II-IV colorectal cancer post-resection.
* Receiving active adjuvant chemotherapy.
* Documented moderate-to-severe malnutrition (PG-SGA score ≥ 4).
* Ability to tolerate oral intake.
* Voluntarily signed the informed consent form.

Exclusion Criteria:

* Presence of complete bowel obstruction.
* Severe, uncontrolled organ dysfunction (cardiac, hepatic, renal).
* Known allergy to any component of the nutritional supplements.
* Concurrent participation in another interventional trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Immunoglobulin A (IgA) level | Baseline and 12 weeks
  Measurement of plasma IgA levels to assess humoral immune response.
Change in Immunoglobulin G (IgG) level | Baseline and 12 weeks
  Measurement of plasma IgG levels to assess humoral immune response.
Change in CD4+/CD8+ T-lymphocyte ratio | Baseline and 12 weeks
  Measurement of the ratio of CD4+ to CD8+ T-lymphocytes from peripheral blood to assess cellular immune status.
Change in Gut Microbiota Alpha Diversity | Baseline and 12 weeks
  Assessment of microbial diversity within fecal samples, measured by the Shannon index based on 16S rRNA gene sequencing.
Change in Relative Abundance of Probiotics | Baseline and 12 weeks
  Quantification of the relative abundance of key probiotic genera (Bifidobacterium, Lactobacillus) in fecal samples via 16S rRNA sequencing.

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline and 12 weeks
  Calculated as weight in kilograms divided by the square of height in meters (kg/m²).
Change in Patient-Generated Subjective Global Assessment (PG-SGA) score | Baseline and 12 weeks
  A validated tool for assessing nutritional status in cancer patients, where lower scores indicate better nutritional status.
Change in Quality of Life (WHOQOL-100) score | Baseline and 12 weeks
  Assessed using the World Health Organization Quality of Life-100 questionnaire, with higher scores indicating better quality of life.
3-Year Overall Survival Rate | Up to 3 years
  Percentage of patients alive at 3 years from the date of study entry.
Incidence of Major Treatment-Related Complications | During the 12-week intervention period
  Number of patients experiencing grade ≥3 complications (e.g., diarrhea, neutropenic fever) during the intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China